CLINICAL TRIAL: NCT03856151
Title: To Evaluate the Effects of Heating Device (Electronic Moxibustion) in Patients With Intradialytic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201801853A3
Record Dates: First submitted 2019-02-11; First posted 2019-02-27 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2019-01

CONDITIONS: Hemodialysis-Induced Symptom; Intra-dialytic Hypotension
Keywords: hemodialysis; Intra-dialytic Hypotension; heating device; electronic moxibustion

STUDY DESIGN:
Intervention Model Description: 30 eligible participants diagnosed with IDH will be enrolled and divided randomly and equally into Group 1 and Group 2 . Treatment 1# will be regular dialysis 3 times per week for 4 weeks. Treatment 2# will be regular dialysis 3 times per week plus "HEALTHY BOX" Powered heating pad on acupoint CV4 at the abdomen for 1 hour during dialysis, also for 4 weeks. For Group 1, each subject will receive Treatment 1# first, for Group 2, Treatment 2# will be received first. Then, a 2-week washout period with regular dialysis 3 times per week will be carried out. Group 1 will then receive Treatment 2# and Group 2 will then receive Treatment 1#. Subjective questionnaires will be done before and after each Treatment period.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): For Group 1, each subject will receive Treatment 1# first. Then, it takes 2-week washout period with regular dialysis 3 times per week and then receive Treatment 2#.
  Treatment 1# will be regular dialysis 3 times per week for 4 weeks. Treatment 2# will be regular dialysis 3 times per week plus "HEALTHY BOX" Powered heating pad on acupoint CV4 at the abdomen for 1 hour during dialysis, also for 4 weeks.
  Interventions: Device: "HEALTHY BOX" Powered heating pad (electronic moxibustion)
- Group 2 (Active Comparator): For Group 2, each subject will receive Treatment 2# first. Then, it takes 2-week washout period with regular dialysis 3 times per week and then receive Treatment 1#.
  Treatment 2# will be regular dialysis 3 times per week plus "HEALTHY BOX" Powered heating pad on acupoint CV4 at the abdomen for 1 hour during dialysis, also for 4 weeks.
  Treatment 1# will be regular dialysis 3 times per week for 4 weeks.
  Interventions: Device: "HEALTHY BOX" Powered heating pad (electronic moxibustion)

INTERVENTIONS:
Device: "HEALTHY BOX" Powered heating pad (electronic moxibustion) — Using heating pad (electronic moxibustion) with insulating materials on low temperatures (56±8℃) in treating patients with intra-dialytic hypotension

SUMMARY:
The aim of this study is to investigate the effects of heating device among otherwise stable patients with intradialytic hypotension

DETAILED DESCRIPTION:
Intradialytic hypotension (IDH) is a common complication during hemodialysis (HD) which accounts up to 5 to 30 percent of all dialysis treatment and is associated with increased morbidity and mortality. The etiology of IDH is multifactorial, but intravascular volume depletion, autonomic neuropathy, and decreased cardiac reserve were the main factors. Several approaches were utilized to prevent IDH including adaptation of dialysis prescriptions, lengthening in dialysis time, avoiding food intake during dialysis, as well as limiting interdialytic sodium intake and administration of vasoconstrictor agents. However, it remains necessary to seek novel effective and safe inventions for IDH. To date, no studies have been done to evaluate the effectiveness of acupuncture and traditional moxibustion during HD for safety reasons (eg: risk of bleeding, burns and unpleasant smell). Therefore, the heating device appears to be a non-invasive and safe method for treating IDH. The investigators conduct a clinical trial using infrared heating devices without direct contact to the skin on low temperatures (56±8℃) in treating patients with IDH. 30 eligible participants diagnosed with IDH will be enrolled and divided into Group 1 and Group 2. Treatment 1# will be regular dialysis 3 times per week for 4 weeks. Treatment 2# will be regular dialysis 3 times per week plus "HEALTHY BOX" Powered heating pad on acupoint CV4 at the abdomen for 1 hour during dialysis, also for 4 weeks. For Group 1, each subject will receive Treatment 1# first, for Group 2, Treatment 2# will be received first. Then, it takes 2-week washout period with regular dialysis 3 times per week and make Group 1 and Group 2 crossover. Outcomes will include blood pressure changes, nursing intervention frequencies, IDH frequencies, the degree of cold intolerance, the degree of fatigue after dialysis and recovery time from fatigue after dialysis, the percentage of target ultrafiltration achieved and blood biochemistry. Data will be collected at the beginning of the study (baseline), end of Treatment 1 # , and end of Treatment 2#. Subjective questionnaires will be collected before and after each treatment period. The difference of evaluation scores between baseline and post-treatment will be analyzed using generalized linear mixed model. A value of P < 0.05 will be regarded as statistically significant for the above statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 80-years-old
2. Willing to sign inform consent
3. Weekly hemodialysis 3 times per week, each time at least 180 minutes
4. During the past 2 months of hemodialysis, there is symptomatic intra-dialytic hypotension for over 15% of the time or under regular use of Midodrine.

Exclusion Criteria:

1. Pregnancy or breast-feeding
2. Not able to fill out questionnaires
3. Severe comorbidities, including cirrhosis, heart failure, autoimmune diseases and cancer
4. Diabetic peripheral neuropathy or patients insensitive to heat or unable to effectively express themselves in heated situations
5. Undergoing other types of alternative treatment, including Chinese medicine and regional remedies.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
change of frequency of IDH episodes | baseline, Treatment 1, Treatment 2
  times of IDH episode according to NADIR, KDOQI criteria
change of number of nursing interventions during HD | baseline, Treatment 1, Treatment 2
  Trendelenburg position, man¬ual reduction of ultrafiltration rate, infusion of isotonic saline or hypertonic fluid, lowering of dialysate temperature

SECONDARY OUTCOMES:
change of the degree of cold intolerance | week 0,4,6,10
  from 0 to 100; 0 is not cold, 100 is very cold
change of the degree of fatigue after dialysis | before and after Treatment1 & 2
  scores from 0-10;0 is not tired, 10 is very tired
blood pressure changes | baseline, Treatment 1, Treatment 2
  systolic, diastolic blood pressure and mean arterial pressure: mmHg
change of recovery time from fatigue after dialysis | before and after Treatment1 & 2
  within minutes (0), when arriving home (0), at bedtime (2), the next morning (5), and by next HD (10)

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No
1. There will be a research number representing the identity. This number will not display the name, ID number, and address.
  2. For the results and diagnosis of the visit, the research host will maintain a confidential attitude and carefully maintain the privacy. If research results are published, the identity will remain confidential.
  3. Please also understand that if the participant signs the consent form, the participant agrees that the visit record can be directly reviewed by the monitor, auditor, research ethics committee and the competent authority to ensure that the research process and data comply with relevant laws and regulations. These people also promise not to violate the confidentiality of your identity.